CLINICAL TRIAL: NCT06796387
Title: SMART-SBAT: Transforming Pediatric Asthma Care Through School-Based Single-Inhaler Therapy
Brief Title: SMART-School-based Asthma Therapy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: Michigan State University (Other)
Responsible Party: Principal Investigator, Jill Halterman, Professor of Pediatrics, Division Director Pediatrics/General, University of Rochester
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00009394
Record Dates: First submitted 2024-05-22; First posted 2025-01-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Asthma in Children

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMART-SBAT (Experimental): In coordination and approval by the child's primary care or specialist provider, children will receive a single maintenance and reliever therapy (SMART) inhaler for school-based asthma therapy (SBAT). Supervised by the school nurse, children will use their prescribed SMART inhaler each school day for preventive therapy, with additional doses as needed to relieve symptoms. Follow-up control assessments will determine if a step-up in therapy may be warranted, and follow-up provider visits will be initiated through school-based telemedicine or in-person visits. An Asthma Coordination team (nurse and community health worker) will be available to coordinate asthma care between providers, pharmacies, schools and families, and provide additional pragmatic support as needed.
  Interventions: Behavioral: SMART-SBAT
- Usual Care (UC) (Active Comparator): Children enrolled in usual care schools will continue to receive asthma management through existing healthcare providers, schools will provide reliever inhalers as prescribed, and preventive asthma therapy is prescribed and delivered through normal channels. Each school year, all school nurses will receive a general orientation on guideline-based asthma management, including SMART and potential benefits of school-based asthma therapy, but standardized workflows or structured coordination will not be available for usual care schools. Caregivers and primary care providers will receive notifications of the child's asthma symptoms and recommendations for SMART therapy.
  Interventions: Behavioral: Usual Care

INTERVENTIONS:
Behavioral: SMART-SBAT — In coordination and approval by the child's primary care or specialist provider, children will receive a single maintenance and reliever therapy (SMART) inhaler for school-based asthma therapy (SBAT). Supervised by the school nurse, children will use their prescribed SMART inhaler each school day for preventive therapy, with additional doses as needed to relieve symptoms. Follow-up control assessments will determine if a step-up in therapy may be warranted, and follow-up provider visits will be initiated through school-based telemedicine or in-person visits. An Asthma Coordination team (nurse and community health worker) will be available to coordinate asthma care between providers, pharmacies, schools and families, and provide additional pragmatic support as needed.
  Arms: SMART-SBAT
Behavioral: Usual Care — Children enrolled in usual care schools will continue to receive asthma management through existing healthcare providers, schools will provide reliever inhalers as prescribed, and preventive asthma therapy is prescribed and delivered through normal channels. Each school year, all school nurses will receive a general orientation on guideline-based asthma management, including SMART and potential benefits of school-based asthma therapy, but standardized workflows or structured coordination will not be available for usual care schools. Caregivers and primary care providers will receive notifications of the child's asthma symptoms and recommendations for SMART therapy.
  Arms: Usual Care (UC)

SUMMARY:
The goal of this research trial is to: 1) Develop a SMART-SBAT protocol specifically designed for schools, 2) Evaluate the effectiveness of SMART-SBAT vs. usual care using a district wide, stepped-wedge type 1 cluster randomized trial and 3) Evaluate the process of implementing SMART-SBAT to contextualize effectiveness outcomes and inform future scale-up.

DETAILED DESCRIPTION:
Despite well-established asthma guidelines and effective preventive medications, many children with persistent asthma do not receive recommended daily anti-inflammatory therapy, and follow-up care with guideline-based step-up adjustments and specialty evaluation is inconsistent. Over a decade ago, in partnership with the Rochester City School District, the investigators co-developed the School-Based Asthma Therapy (SBAT) program to enhance adherence to guideline-based treatment through school-based directly observed therapy (DOT) of preventive medications. Research demonstrated reductions in exacerbations and asthma symptoms, and key stakeholders strongly supported program continuation and scale-up. However, despite its clinical impact, SBAT has not been broadly implemented or sustained outside research trials, and some children continued to have suboptimal asthma control. Recent guideline endorsement of single maintenance and reliever therapy (SMART) offers a timely opportunity to accelerate translation of evidence-based asthma care into real-world practice. SMART simplifies asthma management, improves symptom control, and enables rapid intensification of anti-inflammatory therapy when control remains poor, yet uptake in routine pediatric care remains limited. To address this critical implementation gap and advance pediatric asthma care, the investigators plan to initiate SMART-SBAT, integrating a single ICS-formoterol inhaler at school for both DOT and symptom-driven use. Because school nurses already manage reliever medications, replacing separate controller and reliever inhalers with a single ICS-formoterol inhaler simplifies medication management, facilitates rapid adoption of SMART within existing school health workflows, and enables a "natural" step-up in therapy when symptoms occur. By embedding guideline-recommended SMART delivery in schools, SMART-SBAT provides a pragmatic pathway to accelerate real-world implementation at scale. SMART-SBAT also provides a platform to evaluate treatment response under conditions of reliable medication exposure, including differential effects by asthma phenotype and environmental context, while facilitating specialty evaluation for children with ongoing poor control. Using a pragmatic Type 1 hybrid stepped-wedge trial, the investigators will evaluate effectiveness while simultaneously assessing implementation processes relevant to real-world delivery. Approximately 330 caregivers in SMART-SBAT and usual care schools will be enrolled for longitudinal surveys and medical record reviews to assess outcomes (primary outcome = urgent care and emergency visits for asthma over 12 months). Explanatory mixed-methods analyses will assess reach, fidelity, dose, and adaptations, and evaluate whether baseline clinical characteristics, environmental exposures, and social context modify response to SMART-SBAT. Findings will inform foundational components of a SMART-SBAT toolkit to support broader dissemination. By accelerating uptake of simplified, guideline-based therapy within routine school systems and enabling evaluation beyond adherence barriers, SMART-SBAT aims to reduce exacerbations, improve asthma control, and generate actionable evidence for scalable, high-quality asthma care.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosed asthma, with moderate-severe persistent symptoms or poor control based on NHLBI criteria
* Age >=6 and =<12 years
* Attending school in Rochester City School District
* Caregiver >=18 years, and is able to understand and speak English or Spanish

Exclusion Criteria:

* Caregiver inability to speak and understand English or Spanish. (*Participants unable to read will be eligible, and all instruments will be given verbally.)
* Having other significant medical conditions, including congenital heart disease, cystic fibrosis, or other chronic lung disease, that could interfere with the assessment of asthma-related measures.
* In foster care or other situations in which consent cannot be obtained from a guardian.

Based on prior studies, fewer than 10% of subjects are expected to be excluded based on these criteria.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 330 (Estimated)
Dates: Start 2026-12 (Estimated); Primary Completion 2031-07 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of children with one or more acute health care visits due to asthma over 12 months | 12 months
  The percentage of children who experience one or more acute health care visits (emergency, urgent care) for asthma over 12 months

SECONDARY OUTCOMES:
Mean number of symptom-free days in prior 14 days | 12-month follow-ups
  Mean number of symptom-free days (24 hours without symptoms) in prior 14 days at each follow-up time point (3, 6, 9 and 12 months after baseline).
Mean number of nights with asthma symptoms in prior 2 weeks | 12 months
  Mean number of nights with asthma symptoms in the prior 14 days at each follow-up time point (3, 6, 9 and 12 months after baseline).
Mean number of days requiring use of reliever medication in prior 14 days | 12 months
  Mean number of days requiring reliever therapy in the prior 14 days at each follow-up time point (3, 6, 9 and 12 months after baseline).
Quality of Life Score at 12 months | 12 months
  Pediatric Asthma Caregiver Quality of Life score at each follow-up. Scores range from1-7, higher scores indicate better quality of life.
Asthma Control Score at 12 months | 12 months
  Asthma control score as indicated by the Pediatric Asthma Impairment and Risk Questionnaire (Peds-AIRQ); scores range 0-8; lower scores indicate better asthma control
Number of oral corticosteroid bursts and hospitalizations due to asthma symptoms over 12 months | 12 months
  Total number of oral corticosteroid bursts and hospitalizations over 12 months
FEV1 level | 12 months
  Lung function measured by most recent FEV1 level listed in medical record
Absenteeism due to asthma | 12 months
  Number of days participant misses school due to asthma
Medication Adherence | 12 months
  Caregiver report of missed doses, school medication administration records, Horne Adherence Scale
Program Reach | 12 months
  Proportion of eligible students that enroll into SMART-SBAT
Program Fidelity | 12 months
  Proportion of children where all SMART-SBAT components are delivered (screening, assessment, initiation of SMART-based therapy, and administration of medications in school)
Program Dose | 12 months
  Mean number of program contacts completed per child
Program Adoption | 12 Months
  Proportion of schools reporting readiness and intent to adopt SMART-SBAT with the availability of a standardized toolkit
Program Cost Effectiveness | 12 months
  Evaluation of cost of program per student/participant

IPD SHARING:
Plan to Share IPD: Yes
All raw data produced in the course of the project will be preserved. All de-identified quantitative analysis datasets will be shared once the main study results have been accepted for publication.
  The research data from this project will be deposited within the digital repository of the Inter-university Consortium for Political and Social Research (ICPSR) to ensure that the research community has long-term access to the data, once the main study manuscript has been accepted for publication (or by the end of the grant period; whichever comes first).
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be made available once the results from the main study aims have been accepted for publication or study closure (whichever comes first), and will remain available for 5 years past the grant end date.
Access Criteria: Public-use data files: These files, in which direct and indirect identifiers have been removed to minimize disclosure risk, may be accessed directly through the ICPSR website.
  Restricted-use data files: These files are distributed in those cases when removing potentially identifying information would significantly impair the analytic potential of the data. Users (and their institutions) must request these files from Dr. Halterman and complete a Data Sharing Agreement. The investigator team will review and approve each request.